CLINICAL TRIAL: NCT02380794
Title: Novel Treatment of Intermittent Claudication in Patients With Peripheral Arterial Disease Using Danshen Gegen (D&G) Capsule
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Associated Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DG-PAD
Record Dates: First submitted 2015-02-10; First posted 2015-03-05 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: Danshen Gegen Capsule
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Danshen-Gegen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Danshen Gegen Capsule (Active Comparator): 3 capsules (500 mg per capsule) twice daily for 24 weeks
  Interventions: Drug: Danshen Gegen Capsule
- Placebo (Placebo Comparator): 3 capsules (500 mg per capsule) twice daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Danshen Gegen Capsule — Danshen can dilate blood vessels, reduce the number of angina attacks and significantly improve endothelial function in patients with Coronary Angina Pectoris.
  Gegen is also effective in dilating cardiovascular and cerebrovascular of the brain, and improving blood circulation. The main active ingredient of Gegen isoflavones is effective in dilating the coronary arteries, improving metabolism in normal and ischemic myocardium and reducing blood pressure, heart rate and myocardial oxygen consumption.
  Other Names: D&G
  Arms: Danshen Gegen Capsule
Drug: Placebo
  Arms: Placebo

SUMMARY:
Peripheral arterial disease (PAD) due to lower limb arterial blockages affects significant proportion of the population with an age-adjusted prevalence of approximately 12%. Claudication induced walking impairment can be debilitating and adversely affects social, leisure, and occupational activities in many patients and is associated with higher mortality among PAD patients.

Unfortunately, very few effective therapies are available to improve leg symptoms and exercise performance in PAD patients. Surgery is the last resort but results vary. Therefore, there is a large unmet need for medical therapies that can improve long-term walking performance and functional capacity in PAD patients.

Danshen and Gegen (D&G) are commonly used Chinese herbal medicine in the treatment of cardiovascular diseases. D&G study has been extensively researched and continued at The Chinese University of Hong Kong (CUHK) for their antioxidative and vasodilator properties, modulate anti-atherosclerosis and improve arthrogenic athophysiology. Three randomized trials were completed at the CUHK showing D&G improved lipid profile, vascular function and thinned down the internal layer of the carotid artery. One may expect the same with lower limb arteries. Extensive clinical experiences of use in China and Hong Kong indicated that D&G are well tolerated and safe.

This project is a randomized control trial to determine the efficacy and Safety of D&G in improving the functional capacity & QoL in patients with symptomatic PAD. The results of this study have the potential to change local and international practice in providing a much needed therapeutic option in the treatment of PAD.

DETAILED DESCRIPTION:
Peripheral arterial disease involving the lower limbs is becoming an increasingly important health issue which places considerable burden on individuals, communities and health care resources. PAD affects an estimated 27 million adults >55 years of age in Europe and North America (1). The prevalence of PAD in Asia is expected to be similar and is likely to rise as the Chinese population ages. Intermittent claudication affects most patients with PAD. Although IC is not limb-threatening, the loss of walking ability and the experience of pain with ambulation can cause significant social, leisure, and occupational impairment in many patients (2-4). The decreased QoL experienced in patients with IC is on par with other cardiovascular diseases such as heart failure and heart attack. More alarmingly, physical disability is associated with higher risk of death among PAD patients. For these reasons and because patients are chronically disabled, the treatment of IC has increasingly become a major clinical focus in cardiovascular research.

For PAD patients, it is critical to focus on therapies that can reduce the underlying cardiovascular risk as well as improving functional status and Qol. Although multiple therapies (antiplatelet agents, statins, anti-hypertensive agents) have been proven to reduce cardiovascular risk in PAD patients, very few therapeutic agents have been shown to improve symptoms of IC in PAD patients (5). As such there is a large unmet need in terms of leg-specific therapies that can improve walking performance and functional capacity for this debilitating disease. Traditional Chinese herbal medicine such as Danshen and Gegen are well established in the treatment of cardiovascular diseases and well tolerated by most patients. The studies done at the Institute of Chinese Medicine of the CUHK showed particularly encouraging results (6-8). The outcomes of this study have the potential to change local and international practice in providing a novel therapeutic option in the treatment of symptomatic PAD. As parallel laboratory research is being done to identify the most active components of the D&G formula in preparation for drug development, the efficacy of D&G in PAD will offer more assurance for the systemic efforts.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 40 years or older
2. With stable intermittent claudication secondary to PAD defined as resting ABI <0.90 and a ≥10mmHg decrease in ankle artery blood pressure after exercise.
3. No change in existing therapy for claudication within 3 months of study enrollment.

Exclusion Criteria:

1. Critical limb ischemia defined by ischemic rest pain, ulceration, or gangrene
2. Major lower limb amputation
3. Surgical or endovascular revascularization for PAD within 3 months prior to enrolment
4. Exercise limitation due to significant concomitant disease (e.g. severe arthritis, cardiac or pulmonary disease)
5. Pregnant women and women who are breastfeeding
6. Patients who are currently on Warfarin
7. Patients with resting systolic blood pressure below 100mmHg (SBP < 100mmHg)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Change in total distance walked on a standardized graded treadmill | between baseline and 24 weeks

SECONDARY OUTCOMES:
Change in distance walked to onset of claudication | between baseline and 24 weeks
Change in health related quality of life assessed by EuroQol-5 Dimension | between baseline and 24 weeks
Change in functional status assessed by Walking Impairment Questionnaire | between baseline and 24 weeks
Rates of combined cardiovascular events including vascular death, myocardial infarction, stroke, revascularization, or readmission to hospital for a vascular or atherosclerosis-related complication | At 24 weeks
Change in ankle brachial index before and after exercise by brachial-to-ankle pulse wave velocity | between baseline and 24 weeks
Changes in arterial stiffness assessed by brachial-to-ankle pulse wave velocity | between baseline and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Ping Yen YAN, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

REFERENCES:
- [Background] Criqui MH, Fronek A, Barrett-Connor E, Klauber MR, Gabriel S, Goodman D. The prevalence of peripheral arterial disease in a defined population. Circulation. 1985 Mar;71(3):510-5. doi: 10.1161/01.cir.71.3.510. PMID 3156006
- [Background] Kannel WB, McGee DL. Update on some epidemiologic features of intermittent claudication: the Framingham Study. J Am Geriatr Soc. 1985 Jan;33(1):13-8. doi: 10.1111/j.1532-5415.1985.tb02853.x. PMID 3965550
- [Background] McDermott MM, Greenland P, Liu K, Guralnik JM, Celic L, Criqui MH, Chan C, Martin GJ, Schneider J, Pearce WH, Taylor LM, Clark E. The ankle brachial index is associated with leg function and physical activity: the Walking and Leg Circulation Study. Ann Intern Med. 2002 Jun 18;136(12):873-83. doi: 10.7326/0003-4819-136-12-200206180-00008. PMID 12069561
- [Background] McDermott MM, Liu K, Greenland P, Guralnik JM, Criqui MH, Chan C, Pearce WH, Schneider JR, Ferrucci L, Celic L, Taylor LM, Vonesh E, Martin GJ, Clark E. Functional decline in peripheral arterial disease: associations with the ankle brachial index and leg symptoms. JAMA. 2004 Jul 28;292(4):453-61. doi: 10.1001/jama.292.4.453. PMID 15280343
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 Practice Guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease): endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. Circulation. 2006 Mar 21;113(11):e463-654. doi: 10.1161/CIRCULATIONAHA.106.174526. No abstract available. PMID 16549646
- [Background] Chan YL, Woo KS, Leung PC, Fung KP. Traditional Chinese medicine Danshen-Gegen combination formula improves atherogenic pathophysiology: an in-vitro and ex-vivo study. Journal of the Hong Kong College of Cardiology. 2006;14:28.
- [Background] Tam LWY, Chook, P, Poon PYK, Qiao M, Chan LLT, Cheung ASP, Chan TYK,Fung KP, Tang KSL, Lau VKM, Koon JCM, Leung PC, Celemajer DS, Woo KS. Danshen and Gegen as cardiovascular tonic in coronary patients: a novel strategy for secondary atherosclerosis prevention. Journal of the Hong Kong College of Cardiology. 2004;12:32.
- [Background] McDermott MM, Greenland P, Liu K, Guralnik JM, Criqui MH, Dolan NC, Chan C, Celic L, Pearce WH, Schneider JR, Sharma L, Clark E, Gibson D, Martin GJ. Leg symptoms in peripheral arterial disease: associated clinical characteristics and functional impairment. JAMA. 2001 Oct 3;286(13):1599-606. doi: 10.1001/jama.286.13.1599. PMID 11585483